CLINICAL TRIAL: NCT04240301
Title: Global PRoMiSe (Perioperative Recommendations for Medication Safety): A Consensus-Based, Generalizable Approach
Brief Title: Perioperative Recommendations for Medication Safety
Status: Not yet recruiting | Type: Observational
Sponsor: Karen C. Nanji,M.D.,M.P.H. (Other)
Collaborators: World Federation of Societies of Anesthesiologists (Unknown); University of California, San Francisco (Other); Aga Khan University (Other); University of Toronto (Other); University of Minnesota (Other); University of Auckland, New Zealand (Other)
Responsible Party: Sponsor-Investigator, Karen C. Nanji,M.D.,M.P.H., Assistant Professor of Anesthesia at Harvard Medical School, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Other Study IDs: 2019P003567
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Perioperative Medication Safety
Keywords: medication safety; anesthesiology; perioperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the proposed research is to create and disseminate expert-based recommendations for perioperative medication safety that are tailored to country income level, using the World Bank's four country income groups: high, upper-middle, lower-middle, and low income. The specific aims of the research are to: 1) Develop consensus-based perioperative medication safety recommendations, 2) Prioritize the recommendations by their level of clinical importance for implementation in high, upper-middle, lower-middle and low income countries, and disseminate the recommendations; and 3) Evaluate the initial adoption of the recommendations in each country income group.

DETAILED DESCRIPTION:
The overall objective of the proposed research is to create and disseminate expert-based recommendations for perioperative medication safety that are tailored to country income level, using the World Bank's four country income groups: high, upper-middle, lower-middle, and low income. The proposed project will include the entire medication use process (ordering, dispensing, preparing, administering, documenting and monitoring). The specific aims of the research are to:

1. Develop consensus-based perioperative medication safety recommendations. Approach: This study will use the extensively studied RAND-UCLA Delphi Method to achieve consensus, with an expert panel consisting of anesthesiologists, surgeons, nurses and medication safety experts from each of the World Bank's four country income groups.
2. Prioritize the recommendations by their level of clinical importance for implementation in high, upper-middle, lower-middle and low income countries, and disseminate the recommendations. Approach: The expert panel members will rank each recommendation by its importance as a next step in improving medication safety in each country income group. A Condorcet ranking method will be used to combine individual rankings into a single list of recommendations ranked by the importance of implementation for each country income group. The investigators will then execute a comprehensive dissemination strategy.
3. Evaluate the initial adoption of the recommendations in each country income group. Approach: The investigators will conduct qualitative, one-on-one, semi-structured interviews of the expert panel members, to evaluate their perceptions of initial adoption of the recommendations in each country income group. A grounded theory approach will be used to identify common themes.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologists, surgeons, operating room nurses, nurse anesthetists, pharmacists and patient safety experts

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our expert panel will consist of 120 members, 30 from each of the World Bank's four county country income groups: high, upper-middle, lower-middle, and low income. Expert panel members will be anesthesiologists, surgeons, operating room nurses, nurse anesthetists, pharmacists and patient safety experts.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Expert-based medication safety recommendations. | 3 years
  Four tiers of stepwise recommendations, corresponding to each of the World Bank's four country income groups.

CONTACTS AND LOCATIONS:
Overall Officials: Karen C. Nanji, M.D., M.P.H., Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No
No IPD will be available to other researchers. Aggregate data post-analysis may be shared with collaborators at other institutions.

REFERENCES:
- [Background] Merry AF, Webster CS, Hannam J, Mitchell SJ, Henderson R, Reid P, Edwards KE, Jardim A, Pak N, Cooper J, Hopley L, Frampton C, Short TG. Multimodal system designed to reduce errors in recording and administration of drugs in anaesthesia: prospective randomised clinical evaluation. BMJ. 2011 Sep 22;343:d5543. doi: 10.1136/bmj.d5543. PMID 21940742
- [Background] Nanji KC, Patel A, Shaikh S, Seger DL, Bates DW. Evaluation of Perioperative Medication Errors and Adverse Drug Events. Anesthesiology. 2016 Jan;124(1):25-34. doi: 10.1097/ALN.0000000000000904. PMID 26501385
- [Background] Llewellyn RL, Gordon PC, Wheatcroft D, Lines D, Reed A, Butt AD, Lundgren AC, James MF. Drug administration errors: a prospective survey from three South African teaching hospitals. Anaesth Intensive Care. 2009 Jan;37(1):93-8. doi: 10.1177/0310057X0903700105. PMID 19157353
- [Background] Orser BA, Chen RJ, Yee DA. Medication errors in anesthetic practice: a survey of 687 practitioners. Can J Anaesth. 2001 Feb;48(2):139-46. doi: 10.1007/BF03019726. PMID 11220422
- [Background] Shridhar Iyer U, Fah KK, Chong CK, Macachor J, Chia N. Survey of medication errors among anaesthetists in Singapore. Anaesth Intensive Care. 2011 Nov;39(6):1151-2. No abstract available. PMID 22165377
- [Background] Webster CS, Merry AF, Larsson L, McGrath KA, Weller J. The frequency and nature of drug administration error during anaesthesia. Anaesth Intensive Care. 2001 Oct;29(5):494-500. doi: 10.1177/0310057X0102900508. PMID 11669430
- [Background] Wahr JA, Abernathy JH 3rd, Lazarra EH, Keebler JR, Wall MH, Lynch I, Wolfe R, Cooper RL. Medication safety in the operating room: literature and expert-based recommendations. Br J Anaesth. 2017 Jan;118(1):32-43. doi: 10.1093/bja/aew379. Epub 2016 Dec 30. PMID 28039240
- [Background] Whitaker D, Brattebo G, Trenkler S, Vanags I, Petrini F, Aykac Z, Longrois D, Loer SA, Gaszynski T, Sipylaite J, Copaciu E, Cerny V, Akeson J, Mellin-Olsen J, Abela C, Stecher A, Kozek-Langenecker S, Ratsep I; European Section and Board of Anaesthesiology of the UEMS. The European Board of Anaesthesiology recommendations for safe medication practice: First update. Eur J Anaesthesiol. 2017 Jan;34(1):4-7. doi: 10.1097/EJA.0000000000000531. PMID 27548778
- [Background] Utley M, Gallivan S, Mills M, Mason M, Hargraves C. A consensus process for identifying a prioritised list of study questions. Health Care Manag Sci. 2007 Feb;10(1):105-10. doi: 10.1007/s10729-006-9003-6. PMID 17323658
- [Derived] Nanji KC, Merry AF, Shaikh SD, Pagel C, Deng H, Wahr JA, Gelb AW, Orser BA. Global PRoMiSe (Perioperative Recommendations for Medication Safety): protocol for a mixed-methods study. BMJ Open. 2020 Jun 30;10(6):e038313. doi: 10.1136/bmjopen-2020-038313. PMID 32606066